CLINICAL TRIAL: NCT02750631
Title: Out-patient Wake Therapy, Light Therapy and Sleep Phase Advance for Depression
Acronym: WakeTherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6938
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Unipolar Depression
Keywords: depression; melatonin; light therapy; Wake Therapy; chronobiology
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: All patients receive Chronotherapy, which consists of a night of no sleep ("Wake Therapy") followed by bright lights at their desired sleep time and two nights of Sleep Phase Advance (i.e., sleeping 6 hours earlier than desired for 1 night and 3 hours earlier for the next night, then desired sleep time).
Masking Description: All patients and staff know what the treatment is.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple Therapy (Experimental): Combined Wake Therapy (one night of missed sleep), early morning bright light and sleep phase advance
  Interventions: Other: Triple Therapy

INTERVENTIONS:
Other: Triple Therapy — The intervention consists of three interventions: missing a night of sleep, early morning bright lights and sleep phase advance
  Other Names: Chronotherapeutics

SUMMARY:
Depressed patients miss a night of sleep (Wake Night), then sleep at predetermined times ending at their desired sleep time. Beginning the morning following their Wake Night, patients sit in front of a bright light, continuing morning bright light and specified sleep time for six weeks with weekly visits measuring depressive symptoms.

DETAILED DESCRIPTION:
Nonpsychotic, nonbipolar, physically healthy depressed patients keep sleep, mood and energy logs for a week, complete the Morningness-Eveningness Questionnaire (measuring "morningness" and "eveningness") and determine the time patients want to sleep. Patients then miss a night of sleep and subsequently are allowed later and later sleep times until patients are sleeping at their desired time. Beginning the morning following their Wake Night, patients sit in front of bright lights at their intended wake-up time for the next six weeks and once their allowed sleep time is their intended sleep time, patients also continue to only be allowed to sleep between those times (e.g., 11 p.m. to 7 a.m.). Daily sleep, energy and mood logs and activity monitoring are maintained throughout with weekly clinician ratings. In additional, daily telephone check ins occur during the first week following the Wake Night both to be sure the patient is following the protocol and to obtain symptom ratings. Saliva to be measured for melatonin is collected prior to and following sleep adjustment.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder or persistent depressive disorder or unspecified depressive disorder
* physically healthy
* patients over age 60 need primary care physician's approval, electrocardiogram and Mini Mental Status Examination

Exclusion Criteria:

* medically unstable condition
* bipolar disorder
* current (past six months) substance use disorder
* significant suicide risk
* need for hospitalization
* history of psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression | 1 week
  The Hamilton Rating Scale for Depression is a standard clinician scored rating of depressed mood and the symptoms commonly associated with clinical depression

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Stewart, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
No such plan at present